CLINICAL TRIAL: NCT06430892
Title: Efficacy of the Pressure Optimization Protocol (POP )Versus Conventional Stent Deployment Strategy During Primary Percutaneous Coronary Intervention.
Brief Title: RAPID-POP a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Professor Abdul Hakeem, professor, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-23/2024
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups in 1:1 , one arm will be treated with POP protocol and the other arm will be treated with conventional method.
Who Masked: Outcomes Assessor
Masking Description: This will be an open-label study, however, the outcome assessment will be blinded. A de-identified CD and post-PCI ECG with a unique tracking ID will be evaluated by the team of independent consultants, who will be blinded to the stent placement approach, and primary outcome variables i.e. TIMI flow, slow-flow/no-reflow, and ST-segment resolution will be assessed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POP Protocol (Other): Patients in this arm will be treated according to the POP protocol for stent deployment
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)
- Conventional method (Other): Patients in this arm will be treated with conventional method (rapid inflation-deflation protocol) for stent deployment
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)

INTERVENTIONS:
Procedure: Primary Percutaneous Coronary Intervention (PPCI) — Patients presented with acute myocardial infarction undergoing primary percutaneous coronary intervention with stent deployment

SUMMARY:
Efficacy of the Pressure Optimization Protocol (POP) versus Conventional Stent Deployment Strategy during Primary PCI: An Open Label Randomized Clinical Trial The investigators will compare conventional rapid stent inflation/deflation during primary PCI with higher pressure and prolonged duration of stent deployment

Study Hypothesis: The POP in stent deployment is superior to the conventional stent deployment approach with a significantly higher achievement of the TIMI III flow, significantly lesser occurrence of slow flow/no-reflow, and significantly higher rate of ST-Segment resolution during primary PCI.

DETAILED DESCRIPTION:
Primary Objective The primary objective is to compare the rate of TIMI III flow achievement, slow flow/no-reflow, and ST-segment resolution between POP versus conventional stent deployment strategy during Primary PCI.

Secondary Objective The secondary objective is in-hospital outcome (to compare the rate of major adverse cardiovascular events (MACE) during hospitalization between POP versus conventional stent deployment strategy during Primary PCI.) Material and Methods Study design: An open-label randomized controlled trial (RCT) with blinded outcome assessment Setting: Cath Lab NICVD Karachi ,Hyderabad and Sukkur Duration of study: 6 months Stent Deployment Protocol: Patients will be randomly assigned to either POP or conventional stent deployment approach groups in 1:1 ratio using the block randomization method.

SAMPLE SIZE : 400 patients will be randomized into 2 groups with 1:1 Concealment: Allocation schema will remain accessible to the randomization and allocation team and will be communicated to the screening and recruitment team on a patient-on-patient basis.

Blinding: This will be an open-label study, however, the outcome assessment will be blinded. A de-identified CD and post-PCI ECG with a unique tracking ID will be evaluated by the team of independent consultants, who will be blinded to the stent placement approach, and primary outcome variables i.e. TIMI flow, slow-flow/no-reflow, and ST-segment resolution will be assessed.

Immediately post-procedure, a de-identified CD and post-PCI ECG with a unique tracking ID will be evaluated by the team of independent consultants, who will be blinded to the stent placement approach, and primary outcome variables i.e. TIMI flow, slow-flow/no-reflow, and ST-segment resolution will be assessed. All the patients will be followed at 30 days and incidence of MACE will be recorded.

In order to ensure the integrity and reliability of the data, all procedures and imaging assessments will be carried out by clinicians and technicians trained and standardized in the respective methodologies. Moreover, data will be stored in a secure, electronic database with restricted access to maintain patient confidentiality and data security. Regular data audits will be conducted to ensure accuracy and consistency throughout the trial.

Data Analysis:

Firstly, patient demographics and baseline clinical characteristics will be summarized using means and standard deviations for continuous variables and frequencies with percentages for categorical variables. Kaplan-Meier survival analysis will be used to determine the time-to-event data for outcomes such as target vessel failure, target vessel revascularization, cardiac death, and myocardial infarction. Log-rank tests will be employed to compare survival curves between the POP and Rapid I/D groups. Cox proportional hazards models will be used to compute hazard ratios (HRs) and their 95% confidence intervals (CIs) for each outcome of interest, adjusting for potential confounders.

For categorical outcomes, chi-squared tests or Fisher's exact tests will be used, as appropriate. Continuous outcomes will be assessed using t-tests or Mann-Whitney U tests based on data distribution. Any unmatched or imbalanced variables between the two groups will be controlled using propensity score matching. To address potential confounding factors and biases, a sensitivity analysis will be performed.

Lastly, all statistical analyses will be two-tailed, with a significance level set at p < 0.05. Statistical software such as SPSS or R will be utilized for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* Patients undergoing primary percutaneous coronary intervention (PCI) with stent implantation.
* Presence of significant coronary artery stenosis (greater than 70% diameter reduction) confirmed by angiography.

Exclusion Criteria:

* Patients with Killip class IV
* Patients with significant comorbidities such as end-stage renal disease or advanced liver disease which may interfere with the procedure or follow-up.
* Prior history of coronary artery bypass grafting (CABG).
* Refusal to give consent for study participation or procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
TIMI III flow: TIMI III flow is defined as normal flow with complete filling of the distal vascular bed. | periprocedurally (after stent deployment)
  To assess flow in the vessel after deployment of stent
Slow-flow/no-reflow | periprocedurally (after stent deployment)
  To assess is there any Slow-flow/no-reflow phenomenon , which is TIMI flow grade < 3 and as myocardial blushing grade (MBG) < 2.
ST-segment resolution | Time frame:60minutes after the procedure
  Assessment of ST-segment resolution , The electrocardiographic resolution of the ST-segment elevation is defined as a reduction of > 50% of the ST-segment elevation in the same lead within 60 min after the index procedure

SECONDARY OUTCOMES:
Cardiovascular death ( CV death) | Time frame: during hospitalization (in-hospital)
  cardiovascular death
Myocardial infarction | Time frame: during hospitalization (in-hospital)
  Myocardial infarction of different territory
Stent thrombosis | Time frame: during hospitalization (in-hospital)
  same territory Myocardial infarction
Cerebrovascular accident ( CVA /Stroke) | Time frame: during hospitalization (in-hospital)
  Cerebrovascular events during hospital stay
Arrhythmias | Time frame: during hospitalization (in-hospital)
  Significant arrhythmias requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABDUL HAKEEM, PROF, Principal Investigator — National Institute of Cardiovascular Diseases, Pakistan
Locations (1):
- National institute of cardiovascular diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No